CLINICAL TRIAL: NCT00819351
Title: NOPHO Treatment Protocol for Children (1.0 - 17.9 Years of Age) and Young Adults(18.0-45.0 Years) With Acute Lymphoblastic Leukemia. Intermittent Versus Continuous PEG-asparaginase for Asparagine Depletion
Brief Title: ALL2008 Protocol for Childhood Acute Lymphoblastic Leukemia Intermittent Versus Continuous PEG Asparaginase
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Nordic Society for Pediatric Hematology and Oncology (Other)
Responsible Party: Principal Investigator, Kjeld Schmiegelow, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOPHO ALL2008 PEG Asparaginase
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: acute lymphoblastic leukemia; child; PEG-Asparaginase; EFS; efficacy; childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG-asparaginase 6 weeks intervals (Experimental): PEG-asparaginase (1.000 IU/m2/dose) given at six weeks intervals (from week 13 after diagnosis to week 33).
  All additional therapy (High Dose Methotrexate, Vincristin, Dexamethasone, 6-Mercaptopurine, doxorubicin, intrathecal chemotherapy) is the same in both arms.
  Interventions: Drug: PEG Asparaginase at six weeks interval
- PEG-Asparaginase 2 weeks intervals (Active Comparator): PEG-asparaginase (1.000 IU/m2/dose) given at two weeks intervals (from week 13 after diagnosis to week 33).
  All additional therapy (High Dose Methotrexate, Vincristin, Dexamethasone, 6-Mercaptopurine, doxorubicin, intrathecal chemotherapy) is the same in both arms.
  Interventions: Drug: PEG Asparaginase at two weeks interval

INTERVENTIONS:
Drug: PEG Asparaginase at six weeks interval — PEG-asparaginase (1.000 IU/m2/dose) given at six weeks intervals (until the patient has received 33 weeks of therapy)
  Other Names: Oncaspar (PEG-Asparaginase)
  Arms: PEG-asparaginase 6 weeks intervals
Drug: PEG Asparaginase at two weeks interval — PEG-asparaginase (1.000 IU/m2/dose) given at two weeks intervals (until the patient has received 33 weeks of therapy)
  Other Names: Oncaspar (PEG-Asparaginase)
  Arms: PEG-Asparaginase 2 weeks intervals

SUMMARY:
The purpose of this study is to investigate if intramuscular PEG-asparaginase administered either at six or two week intervals from day 92 until 8 months from diagnosis for patients with non-HR ALL will result in equal probability of Event Free Survival

DETAILED DESCRIPTION:
20% of children with ALL still fails to be cured. The ALL-2008 protocol is a treatment and research protocol that aims to improve the overall outcome of Nordic children and adolescents with ALL in comparison with the ALL-2000 protocol and previous NOPHO protocols.

The specific and primary objectives of the randomised study is:

To test if intramuscular PEG-asparaginase administered either at six or two week intervals from day 92 until 8 months from diagnosis for patients with non-HR ALL will result in equal probability of EFS. As secondary endpoints asparaginase antibody production and toxicity including allergic reactions in the treatment-arms will be analysed

ELIGIBILITY:
Inclusion Criteria:

* Childhood ALL
* All mandatory biological data are available6
* Written informed consent has been obtained

Exclusion Criteria:

* Bilineage ALL
* Pre-treatment with glucocorticosteroids or other antileukemic agents for more than 1 week
* ALL predisposition syndromes
* Previous cancer
* Off protocol administration of additional chemotherapy during induction therapy
* Sexually active females not using contraception
* No allergic reactions to PEG Asparaginase

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 650 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2016-03-02 (Actual); Study Completion 2016-03-02 (Actual)

PRIMARY OUTCOMES:
Event Free Survival | 6 years

SECONDARY OUTCOMES:
Secondary Outcome Measures are toxicity (special focus on thrombosis, pancreatitis, and allergic reactions), the formation of silent antibodies, and the influence of antibody production on the EFS. | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Schmiegelow, M.D., Study Chair — Rigshospitalet, Blegdamsvej 9, 2100 Copenhagen
Locations (6):
- Department of Pediatrics, Rigshospitalet, Copenhagen, Denmark
- Helsinki University Hospital, Helsinki, Finland
- University Hospital Reykjavik, Iceland, Reykjavik, Iceland
- Trondheim University Hospital, Trondheim, Norway
- Sweden (2):
  - Department of Pediatrics, Drottning Sylvias Pediatric Hospital, Gothenburg
  - NOPHO nordic organisation for pediatric onology, Stockholm

REFERENCES:
- [Derived] Albertsen BK, Grell K, Abrahamsson J, Lund B, Vettenranta K, Jonsson OG, Frandsen TL, Wolthers BO, Heyman M, Schmiegelow K. Intermittent Versus Continuous PEG-Asparaginase to Reduce Asparaginase-Associated Toxicities: A NOPHO ALL2008 Randomized Study. J Clin Oncol. 2019 Jul 1;37(19):1638-1646. doi: 10.1200/JCO.18.01877. Epub 2019 Apr 12. PMID 30978155
- [Derived] Tram Henriksen L, Gottschalk Hojfeldt S, Schmiegelow K, Frandsen TL, Skov Wehner P, Schroder H, Klug Albertsen B; Nordic Society of Pediatric Hematology and Oncology, NOPHO Group. Prolonged first-line PEG-asparaginase treatment in pediatric acute lymphoblastic leukemia in the NOPHO ALL2008 protocol-Pharmacokinetics and antibody formation. Pediatr Blood Cancer. 2017 Dec;64(12). doi: 10.1002/pbc.26686. Epub 2017 Jun 29. PMID 28660740
- [Derived] Nielsen SN, Grell K, Nersting J, Abrahamsson J, Lund B, Kanerva J, Jonsson OG, Vaitkeviciene G, Pruunsild K, Hjalgrim LL, Schmiegelow K. DNA-thioguanine nucleotide concentration and relapse-free survival during maintenance therapy of childhood acute lymphoblastic leukaemia (NOPHO ALL2008): a prospective substudy of a phase 3 trial. Lancet Oncol. 2017 Apr;18(4):515-524. doi: 10.1016/S1470-2045(17)30154-7. Epub 2017 Mar 1. PMID 28258828
- [Derived] Wolthers BO, Frandsen TL, Abrahamsson J, Albertsen BK, Helt LR, Heyman M, Jonsson OG, Korgvee LT, Lund B, Raja RA, Rasmussen KK, Taskinen M, Tulstrup M, Vaitkeviciene GE, Yadav R, Gupta R, Schmiegelow K. Asparaginase-associated pancreatitis: a study on phenotype and genotype in the NOPHO ALL2008 protocol. Leukemia. 2017 Feb;31(2):325-332. doi: 10.1038/leu.2016.203. Epub 2016 Jul 25. PMID 27451978
- [Derived] Henriksen LT, Harila-Saari A, Ruud E, Abrahamsson J, Pruunsild K, Vaitkeviciene G, Jonsson OG, Schmiegelow K, Heyman M, Schroder H, Albertsen BK; Nordic Society of Paediatric Haematology and Oncology (NOPHO) group. PEG-asparaginase allergy in children with acute lymphoblastic leukemia in the NOPHO ALL2008 protocol. Pediatr Blood Cancer. 2015 Mar;62(3):427-33. doi: 10.1002/pbc.25319. Epub 2014 Nov 21. PMID 25418987
- [Derived] Raja RA, Schmiegelow K, Albertsen BK, Prunsild K, Zeller B, Vaitkeviciene G, Abrahamsson J, Heyman M, Taskinen M, Harila-Saari A, Kanerva J, Frandsen TL; Nordic Society of Paediatric Haematology and Oncology (NOPHO) group. Asparaginase-associated pancreatitis in children with acute lymphoblastic leukaemia in the NOPHO ALL2008 protocol. Br J Haematol. 2014 Apr;165(1):126-33. doi: 10.1111/bjh.12733. Epub 2014 Jan 15. PMID 24428625